CLINICAL TRIAL: NCT01925872
Title: The Optimal Regimen of Medical Treatment in Endovascular Therapy in Ischemic Cerebrovascular Disease Based on Clopidogrel Resistance
Brief Title: Optimal Regimen in Endovascular Therapy in Ischemic Cerebrovascular Disease Based on Clopidogrel Resistance
Acronym: ORETCR
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Zhongrong Miao (Other)
Responsible Party: Sponsor-Investigator, Zhongrong Miao, principal investigator, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Other Study IDs: BTH-GENE-CR
Record Dates: First submitted 2013-08-15; First posted 2013-08-20 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2013-08

CONDITIONS: Ischemic Cerebrovascular Disease
Keywords: ischemic cerebrovascular disease; Percutaneous transluminal angioplasty and stenting; Clopidogrel resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood were retained to extract DNA for genetic sequencing.
Oversight: Data Monitoring Committee: No

SUMMARY:
1. Clopidogrel resistance is common in patients of ischemic cerebrovascular disease.
2. Genetic polymorphisms are the most important factors to clopidogrel resistance.
3. The purpose of this study is to find the genes which are the related to clopidogrel resistance.
4. Through gene sequencing, we can filter patient of clopidogrel resistance, so another drug maybe used to avoid the undesired efficacy.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic ischemic cerebrovascular disease caused by Intracranial atherosclerotic atherosclerosis research database.
* 90 days had a stroke or transient ischemic attack is defined as symptomatic Intracranial atherosclerotic atherosclerosis
* stenosis ≥ 50% (MRI or CT angiography).
* Intracranial vascular stenosis measured according to the method reported Warfarin aspirin symptomatic intracranial disease research.

Exclusion Criteria:

* diffuse intracranial arterial stenosis.
* cranial magnetic resonance imaging shows lesions as the branch artery blockage caused.
* non-atherosclerotic lesions.
* occurred within 6 weeks of vascular lesions in the region of intracranial hemorrhage.
* potential cardiac thrombus source.
* has concurrent intracranial tumors, intracranial aneurysm or arteriovenous malformation.
* ipsilateral extracranial carotid or vertebral artery stenosis ≥ 50%;
* known to heparin, aspirin, clopidogrel, anesthetics and contrast agents contraindications;
* hemoglobin less than 10g/dL, platelet count <100000/dL;
* responsibility left after cerebral vascular-related serious neurological dysfunction (mRS ≥ 3);
* international normalized ratio> 1.5
* there are factors that can not be corrected by bleeding;
* life expectancy <1 year;
* pregnant or lactating women;
* indications Commission determines that the patient is not suitable for the study treatment.

Ages: 25 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic ischemic cerebrovascular disease caused by Intracranial atherosclerotic atherosclerosis research database; 90 days had a stroke or TIA is defined as symptomatic Intracranial atherosclerotic atherosclerosis; Stenosis ≥ 50% (MRI or CT angiography); Intracranial vascular stenosis measured according to the method reported Warfarin aspirin symptomatic intracranial disease research.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
genotype, platelet aggregation rate, cerebrovascular events | 2 years
  Genotype means the genetic polymorphism of ABCB1, CES, CYP2C19, PON1, P2RY12, which can be determined through gene sequencing.

SECONDARY OUTCOMES:
Active metabolite concentration | 2 years
  Active metabolite concentration depend on the genetic polymorphism.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Ma, Doctor, Study Director — Beijing Tiantan Hospital

REFERENCES:
- [Derived] Li XG, Ma N, Sun SS, Xu Z, Li W, Wang YJ, Yang X, Miao ZR, Zhao ZG. Association of genetic variant and platelet function in patients undergoing neuroendovascular stenting. Postgrad Med J. 2017 Sep;93(1103):555-559. doi: 10.1136/postgradmedj-2016-134745. Epub 2017 Mar 9. PMID 28280103
- [Derived] Wang B, Li XQ, Ma N, Mo D, Gao F, Sun X, Xu X, Liu L, Song L, Li XG, Zhao Z, Zhao X, Miao ZR. Association of thrombelastographic parameters with post-stenting ischemic events. J Neurointerv Surg. 2017 Feb;9(2):192-195. doi: 10.1136/neurintsurg-2015-011687. Epub 2015 Jun 3. PMID 26041100